CLINICAL TRIAL: NCT01631487
Title: A Double-Blind, Randomized, Placebo-Controlled, Sequential Group, Single Ascending and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-39439335 in Healthy Japanese and Caucasian Adult Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-39439335 in Healthy Japanese and Caucasian Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100890; 39439335PAI1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; JNJ-39439335; Japanese; Caucasian; Male

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- Japanese Group 1: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 10 mg; Drug: Placebo
- Japanese Group 2: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 25 mg; Drug: Placebo
- Japanese Group 3: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 50 mg; Drug: Placebo
- Caucasian Group 1: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 10 mg; Drug: Placebo
- Caucasian Group 2: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 25 mg; Drug: Placebo
- Caucasian Group 3: JNJ-39439335/placebo (Part 1) (Experimental)
  Interventions: Drug: JNJ-39439335 50 mg; Drug: Placebo
- Japanese Group 1: JNJ-39439335/placebo (Part 2) (Experimental)
  Interventions: Drug: JNJ-39439335 10 mg; Drug: Placebo
- Japanese Group 2: JNJ-39439335/placebo (Part 2) (Experimental)
  Interventions: Drug: JNJ-39439335 25 mg; Drug: Placebo
- Japanese Group 3: JNJ-39439335/placebo (Part 2) (Experimental)
  Interventions: Drug: JNJ-39439335 50 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-39439335 10 mg — Multiple (once daily for 21 days) oral doses of JNJ-39439335 10 mg.
  Arms: Caucasian Group 1: JNJ-39439335/placebo (Part 1); Japanese Group 1: JNJ-39439335/placebo (Part 1); Japanese Group 1: JNJ-39439335/placebo (Part 2)
Drug: JNJ-39439335 25 mg — Multiple (once daily for 21 days) oral doses of JNJ-39439335 25 mg.
  Arms: Caucasian Group 2: JNJ-39439335/placebo (Part 1); Japanese Group 2: JNJ-39439335/placebo (Part 1); Japanese Group 2: JNJ-39439335/placebo (Part 2)
Drug: JNJ-39439335 50 mg — Multiple (once daily for 21 days) oral doses of JNJ-39439335 50 mg.
  Arms: Caucasian Group 3: JNJ-39439335/placebo (Part 1); Japanese Group 3: JNJ-39439335/placebo (Part 1); Japanese Group 3: JNJ-39439335/placebo (Part 2)
Drug: Placebo — Multiple (once daily for 21 days) oral doses of matching placebo.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of JNJ-39439335 in healthy Japanese and Caucasian adult male participants in Part 1, and in healthy Japanese adult male participants in Part 2.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), randomized (the study drug is assigned by chance), placebo-controlled study (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial). The study consists of 2 Parts. In Part 1, three groups of healthy Japanese men and 3 groups of healthy Caucasian men will receive a single oral dose of JNJ-39439335 or placebo on Day 1. Each group will include 8 participants. The study duration of Part 1 for each participant is approximately 8 weeks: screening phase of up to 28 days prior to dose, treatment phase of 14 days, and a follow-up phase of 14 to16 days. In Part 2, three groups of healthy Japanese men will receive once-daily doses of either JNJ-39439335 or placebo for 21 days. Each group will include 12 participants. The study duration of Part 2 for each participant is approximately 11 weeks: screening phase of up to 28 days prior to dose, treatment phase of 21 days, and a follow-up phase of approximately 28 days. During the treatment phases, the participants will remain in the study unit. Blood samples and urine will be collected for drug concentration measurements and laboratory safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Japanese or Caucasian participants
* Nonsmoker
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive, and body weight not less than 50 kg
* Healthy on the basis of a physical examination, vital signs, hematology, coagulation, serum chemistry (including liver function tests) and urinalysis
* Willing to adhere to the prohibitions and restrictions specified by the study protocol

Exclusion Criteria:

* Oral temperatures > 37.5 Celsius degrees
* Participants who have occupations or hobbies in which they are routinely exposed to situations in which they could sustain thermal burns
* Abnormal electrocardiogram (ECG) results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis
* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of JNJ-39439335 (Part 1) | up to 14 days
Urine concentrations of JNJ-39439335 (Part 1) | up to 5 days
Plasma concentrations of JNJ-39439335 (Part 2) | up to 21 days
Urine concentrations of JNJ-39439335 (Part 2) | up to 21 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (Part 1) | Approximately 8 weeks
Incidence of Adverse Events (Part 2) | Approximately 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States